CLINICAL TRIAL: NCT01679379
Title: Surgical Site Infection in Obese Women After Cesarean Section; A Randomized Controlled Trial of Absorbable Versus Non Absorbable Sutures for Skin Closure.
Brief Title: Wound Infection in Obese Women After Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Ellaithy, Lecturer of Obstetrics & Gynecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ASU-07-2012
Record Dates: First submitted 2012-09-03; First posted 2012-09-06 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Surgical Site Infection
Keywords: Cesarean Section; Obese Women; Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Absorbable suture group (Active Comparator): Include women who have their skin closed with subcuticular stitches using [Polyglactin 910 absorbable, synthetic, braided suture].
  Interventions: Procedure: Absorbable suture group
- Non absorbable suture group (Active Comparator): Include women who have their skin closed with subcuticular stitches using [Polypropylene non absorbable monofilament suture].
  Interventions: Procedure: Non absorbable suture group

INTERVENTIONS:
Procedure: Absorbable suture group — Skin is closed with subcuticular stitches using [Polyglactin 910 absorbable, synthetic, braided suture]
  Arms: Absorbable suture group
Procedure: Non absorbable suture group — Skin is closed with subcuticular stitches using Polypropylene non absorbable monofilament suture
  Arms: Non absorbable suture group

SUMMARY:
The purpose of this study is to determine the surgical site infection rate and patient satisfaction for absorbable versus non absorbable suture in closure of skin at cesarean section in obese women.

DETAILED DESCRIPTION:
Cesarean section (CS) is the commonest major operation performed on women in the world. Approximately one in 4 women in the United States is delivered by cesarean section, and it is well established that operative abdominal delivery is associated with a significant risk of infection compared with vaginal delivery. These risks are increased with preexisting operative site infection, breaks in sterile technique, prolonged preoperative admissions that may result in colonization with resistant microbes, prolonged operative duration, use of electrocautery, obesity, advanced age, inadequate host immunocompetence.

Obese women may have increased susceptibility to infections because of the effects of obesity on the immune system, skin barriers, wound healing, mobility, and coexisting chronic diseases including diabetes, which could increase infection risk by itself. Cohort studies have shown that women with a body mass index (BMI)>30kg/m^2 have a two to three folds increased risk of post cesarean infections, such as wound infection, urinary tract infection UTI), endometritis, or pneumonia, compared with non-obese women. Other studies found that obesity doubled the risk specifically for post-cesarean wound infection.

Wound complications are a major source of morbidity after CS and contribute to prolonged hospital stay and rates of readmission. Age, (BMI), length of incision, and timing of prophylactic antibiotic administration have all been associated with post cesarean surgical site infection (SSI).

A surgical site infection is an infection that occurs after surgery in the part of the body where the surgery took place. SSI can sometimes be superficial infections involving the skin only. Other surgical site infections are more serious and can involve tissues under the skin, organs, or implanted material. SSI has a great impact on the economy and health care resources. Infection has always been a feature of modern surgery and continues to be a significant problem for health care practitioners across the world.

The ideal skin closure would be safe and effective, associated with minimal patient discomfort, and have a good cosmetic result. It would also be inexpensive and require fewer health care resources by being fast and easy to apply, require minimal follow-up evaluation, and be associated with a low rate of complications.

Methods for closing the skin at the time of cesarean delivery include stainless steel staples, subcuticular absorbable staples, subcuticular suture, adhesive closure strips, and tissue adhesives (cyanoacrylates). Each of the methods has its postulated benefits for wound outcomes; however, none of these have been compared in a prospective trial.

The role of skin closure suture material on wound complication rates in Obstetrics is poorly studied. And when we are talking about obese patients we did not find any recommendation regarding the suture material of skin closure although most of Obstetricians use different sutures materials.

Does closure of skin by absorbable compared to non absorbable suture affect the rate of surgical site infection in obese patients undergoing caesarian section? Our hypothesis is that no difference between absorbable compared to non absorbable suture.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant female in child bearing period
* Mode of delivery is by cesarean section (CS)
* Obese women, Body Mass Index (BMI) >30kg/m^2
* Viable fetus
* Gestational age >34 weeks

Exclusion Criteria:

* Hemoglobin (Hb)less than 10g/dl.
* Previous laparotomy other than CS.
* Rupture of membranes for more than 12 hours.
* Presence of signs of systemic or local infection on admission (e.g. fever, tender uterus).
* Prolonged operative time >90 minutes.
* Previous two CS or more.
* Autoimmune disease.
* Immune suppressive disease.
* Corticosteroid medications.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2012-07; Primary Completion 2013-04 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | Within 30 days of surgery
  Diagnosis consists of infection of an anatomic plane by one of the following manifestations: collection; inflammatory signs (pain, tenderness, edema, redness); dehiscence(Wound separation was defined as any separation of the wound that was identified as such by the patient or the medical record and varied in size from small skin defects to separation of the entire wound; or positive culture.

SECONDARY OUTCOMES:
Skin closure time | 30 days
  Complete wound closure

OTHER OUTCOMES:
Postoperative pain | 7 Days
  Women specify their pain level according to visual analogue scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Gamal F. Mostafa, MD, Study Director — Assistant Professor of Obstetrics & Gynecology Faculty of Medicine, Ain Shams University
Locations (1):
- Ain shams university, Cairo, Egypt